CLINICAL TRIAL: NCT04124107
Title: Diagnostic Performance of 68Ga-PSMA PET/MRI in Suspicious Biopsy-naive Prostate Cancer Patients With Favorable Lesion on PET But Unfavorable on MRI for Primary Prostate Cancer Detection: a Pilot Study
Brief Title: Unfavorable MRI But Favorable 68Ga-PSMA PET/MRI for Primary Prostate Cancer Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET+/MRI- v1.0 20191010
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate biopsy with 68Ga-PSMA PET/MRI (Experimental): Both targeted biopsy and 12-core systematic biopsy with positive 68Ga-PSMA PET/MRI
  Interventions: Device: multiparametric MRI and 68Ga-PSMA PET/MRI; Procedure: Prostate biopsy

INTERVENTIONS:
Device: multiparametric MRI and 68Ga-PSMA PET/MRI — All participants will undergo multiparametric MRI examination. If mpMRI is unfavorable for prostate cancer, participants will undergo 68Ga-PSMA PET/MRI examination
Procedure: Prostate biopsy — Participants with unfavorable mpMRI but favorable 68Ga-PSMA PET/MRI will undergo both 68Ga-PSMA PET/MRI-ultrasound-fusion targeted biopsy and transperineal ultrasound guided 12-core systematic biopsy

SUMMARY:
This perspective cohort study aims to assess the detection rate of prostate cancer through prostate biopsy within suspicious patients harboring unfavorable multiparametric MRI but favorable 68Ga-PSMA PET/MRI who have had no prior prostate biopsy.

DETAILED DESCRIPTION:
Multiparametric MRI (MpMRI) is currently regarded as the best imaging method to noninvasively identify and characterize prostate cancer (PCa) with the Prostate Imaging Reporting and Data System (PI-RADS) v2. However, there are diagnostic difficulties for suspicious patients with PI-RADS score 3 and not all PCa are equivalently visible on mpMRI. For such patients, other alternative imaging techniques are required to properly characterize and detect PCa.

It has been widely reported that 68Ga-PSMA PET imaging offers excellent performance in detecting primary PCa and is able to noninvasively characterize the aggressiveness of PCa. Recently, integrated PET/MRI, which combines the strengths of both modalities, has been shown to have great potential for influencing clinical practice by providing a more certain map of localized PCa to aid targeted biopsies and therapy.

This perspective cohort study aims to assess the detection rate of PCa through prostate biopsy within suspicious patients harboring unfavorable mpMRI but favorable 68Ga-PSMA PET/MRI who have had no prior prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Men more than 18 years old with clinical suspicion of prostate cancer;
2. Serum prostate-specific antigen (PSA) > 4 ng/ml within the previous 3 months;
3. PI-RADS score no more than 3 or normal mpMRI of prostate;
4. Suspicious lesion(s) within prostate on 68Ga-PSMA PET/MRI;
5. no evidence of PSA increase by noncancerous factors, such as catheterization, bladder stones, or urinary tract infection including bacterial prostatitis;
6. Able to provide written informed consent.

Exclusion Criteria:

1. Prior prostate biopsy or prostate surgery;
2. Prior treatment for prostate cancer;
3. Contraindication to MRI or PET (e.g. claustrophobia, pacemaker, estimated glomerular filtration rate ≤ 50mls/min);
4. Contraindication to prostate biopsy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of prostate cancer | 30 days post biopsy
  Detection rate of prostate cancer

SECONDARY OUTCOMES:
Detection rates of clinically significant PCa and clinically insignificant prostate cancer | 30 days post biopsy
  Detection rates of clinically significant PCa and clinically insignificant prostate cancer
Gleason grade group distribution (score from 1 to 5, the bigger the score, the worse the prognosis) and aggressive architecture (such as cribriform) on final pathology | 90 days post biopsy
  Gleason grade group distribution (score from 1 to 5, the bigger the score, the worse the prognosis) and aggressive architecture (such as cribriform) on final pathology
Optimal cut-off uptake value on PET/MRI for prostate cancer detection | 30 days post-biopsy
  Optimal cut-off uptake value on PET/MRI for prostate cancer detection

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, PhD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School